CLINICAL TRIAL: NCT05884008
Title: Coronary Computed Tomography Angiography and Functional Analysis in Risk Stratification of Coronary Artery Disease: A Retrospective Cohort Study
Brief Title: Risk Evaluation by COronary CTA and Artificial intelliGence Based fuNctIonal analyZing tEchniques - I
Acronym: RECOGNIZE-I
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Director of Cardiology Department, Principal Investigator, Ruijin Hospital
Other Study IDs: 2022YFC2533502-1
Record Dates: First submitted 2023-05-04; First posted 2023-06-01 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary CTA; CT-FFR; Artificial Intelligence; Risk Stratification
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter, retrospective imaging study. The study intends to retrospectively enroll patients with acute myocardial infarction who had received coronary CTA in a certain time-window before this event. All coronary CTA will be analyzed by anatomic, functional and radiomic analysis, assisted by artificial intelligence. The purpose of this study is to establish a coronary artery disease risk stratification system by coronary CTA.

DETAILED DESCRIPTION:
Coronary angiography has been the gold standard for the diagnosis of coronary heart disease and PCI decision-making. However, the value of CAG in risk stratification is limited due to its invasive nature and lack of ability to evaluate coronary physiology and plaque characteristics, which often leads to over-treatment or under-treatment. In recent years, with the development and improvement of imaging technology, the resolution and diagnostic accuracy of coronary artery CTA have been greatly improved, and the subsequent anatomy and function (non-invasive CT-FFR, etc.) have made the assessment of coronary artery lesion risk multi-dimensional. Comprehensive and accurate coronary artery CTA scan plays a positive role in establishing the appropriate standard for PCI and improving the prognosis of patients. However, the existing problems of coronary artery CTA are insufficient imaging studies, complex image analysis, inconsistent diagnostic criteria, and insufficient clinical evidence. This study is one of the series of clinical studies on the topic of "Risk Evaluation by COronary Computed Tomography and Artificial Intelligence Based fuNctIonal analyZing tEchniques (RECOGNIZE)". The purpose of the study is to establish a coronary artery disease risk stratification system by coronary CTA and anatomic, functional and radiomic analysis, assisted by artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old
* Received coronary CT angiography 3 months to 5 years prior to acute coronary myocardial infarction. CCTA identified coronary atherosclerotic plaques with diameter stenosis ≥ 10%

Exclusion Criteria:

* Familial hypercholesterolemia
* Prior history of percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Prior history of myocardial infarction before the recent event
* Severe liver or renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective imaging study. Clinical records and image of patients received coronary CT angiography 3 months to 5 years prior to acute coronary myocardial infarction from nine clinical centers across P.R. China will be gathered.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary artery plaque risk level | 3 months to 5 years prior to acute myocardial infarction
  Coronary plaque risk was determined using an artificial intelligence (AI) guided risk stratification model based on Coronary CTA structural, functional and radiomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, M.D., Ph.D., Principal Investigator — Ruijin Hospital; Lin Lu, M.D., Ph.D., Study Chair — Ruijin Hospital
Locations (9):
- China (9):
  - Cangzhou Center Hospital, Cangzhou, Hebei
  - First affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - First affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Techonology, Wuhan, Hubei
  - First Hospital of Nanjing, Nanjing, Jiangsu
  - First affiliated hospital of Dalian Medical College, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided